CLINICAL TRIAL: NCT00728468
Title: A Phase 1 Open Label, Single Arm Trial To Evaluate The Effect Of Pf-00299804 On The Pharmacokinetics Of Dextromethorphan In Patients With Advanced Malignant Solid Tumors
Brief Title: A Study To Test The Impact Of PF- 00299804 On How The Body Handles Dextromethorphan In Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Roswell Park Cancer Institute (Other); South Texas Accelerated Research Therapeutics (START) (Unknown)
Responsible Party: Sponsor
Masking: None
Other Study IDs: A7471014
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: Phase 1; PF-00299804; Dextromethorphan; CYP2D6 Inhibition; Cancer Patients
MeSH Terms: interventions — dacomitinib

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — PF-00299804: Patients take oral 45 mg PF-00299804 once daily starting on Cycle 1 Day 1 until disease progression or unacceptable toxicities occur. One cycle equals 21 days. Dextromethorphan: Patient take a single 30 mg oral dose of dextromethorphan HBr three days prior to Cycle 1 Day 1, and then on Cycle 2 Day 7.

SUMMARY:
Research in test tubes suggests that may affect cytochrome P450 2D6 (CYP2D6), an important enzyme that is responsible for eliminating many drugs that cancer patients need to take, including dextromethorphan. The purpose of this study is to test the impact of PF-00299804 on the activity of CYP2D6, and how the human body handles dextromethorphan.

DETAILED DESCRIPTION:
To assess the effect of repeated dosing with 45 mg QD PF-00299804 on the pharmacokinetics of dextromethorphan, a CYP2D6 probe, in cancer patients with advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically or cytologically confirmed advanced malignant solid tumor for which there is no currently approved treatment or which is unresponsive to currently approved therapies;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1. Patients with performance status 2 could be eligible upon agreement between sponsors and investigators;
* Adequate bone marrow, renal, liver and cardiac functions;

Exclusion Criteria:

* History of Interstitial Lung Disease (ILD).
* Drugs with known CYP2D6 inhibitory effects
* Drugs that are highly dependent on CYP2D6 for metabolism.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471014&StudyName=A%20Study%20To%20Test%20The%20Impact%20Of%20PF-%2000299804%20On%20How%20The%20Body%20Handles%20Dextromethorphan%20In%20Cancer%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-00299804 45 mg + Dextromethorphan 30 mg: PF-00299804 45 milligram (mg) tablet orally once daily, starting from Cycle 1 Day 1, continuously for 21-day cycles until disease progression or unacceptable toxicities along with single dose of dextromethorphan hydrobromide 30 mg orally 3 days prior to Cycle 1 Day 1 (Day -3) and on Day 7 of Cycle 2.
Period: Overall Study
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Started | 16
Treated | 15
Completed | 0
Not Completed | 16
Not completed — Enrolled but not treated | 1
Not completed — Death | 1
Not completed — Protocol Violation | 4
Not completed — Objective progression or relapse | 9
Not completed — Study terminated by sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) For Dextromethorphan and Dextrorphan 3 Days Prior to PF-00299804 Dosing
Description: Area under the plasma concentration time-curve from time zero (pre-dose) to the last measured concentration (AUClast). Dextrorphan is an active metabolite of dextromethorphan.
Time Frame: Day -3: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: Pharmacokinetic (PK) analysis population included all participants that were extensive metabolizers and treated, had at least 1 of PK parameters of primary interest in at least 1 treatment period. Here, N (number of participants analyzed) signifies who received PF-00299804 daily without interruptions or dose reductions prior to Day 7 of Cycle 2.
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
nanograms*hour/milliliter (ng*hr/mL)
  Dextromethorphan | 206.4 (404.63)
  Dextrorphan | 2199 (1085.7)

2. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) For Dextromethorphan and Dextrorphan on Cycle 2 Day 7
Description: as for outcome 1
Time Frame: Cycle 2 Day 7: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: PK analysis population included all participants that were extensive metabolizers and treated, had at least 1 of PK parameters of primary interest in at least 1 treatment period. Here, N (number of participants analyzed) signifies who received PF-00299804 daily without interruptions or dose reductions prior to Day 7 of Cycle 2.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
ng*hr/mL
  Dextromethorphan | 300.7 (408.42)
  Dextrorphan | 2232 (1253.2)

3. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) For Dextrorphan 3 Days Prior to PF-00299804 Dosing
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf). Dextrorphan is an active metabolite of dextromethorphan.
Time Frame: Day -3: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
ng*hr/mL | 2266 (955.97)

4. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) For Dextrorphan on Cycle 2 Day 7
Description: as for outcome 3
Time Frame: Cycle 2 Day 7: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
ng*hr/mL | 2298 (1245.4)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) For Dextromethorphan and Dextrorphan 3 Days Prior to PF-00299804 Dosing
Description: Dextrorphan is an active metabolite of dextromethorphan.
Time Frame: Day -3: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
ng/mL
  Dextromethorphan | 6.598 (7.4826)
  Dextrorphan | 239.2 (137.56)

6. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) For Dextromethorphan and Dextrorphan on Cycle 2 Day 7
Description: Dextrorphan is an active metabolite of dextromethorphan.
Time Frame: Cycle 2 Day 7: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
ng/mL
  Dextromethorphan | 11.11 (7.8689)
  Dextrorphan | 169.2 (103.18)

7. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) For Dextromethorphan and Dextrorphan 3 Days Prior to PF-00299804 Dosing
Description: Dextrorphan is an active metabolite of dextromethorphan.
Time Frame: Day -3: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
hours
  Dextromethorphan | 2.00 [1.03 to 6.00]
  Dextrorphan | 2.00 [2.00 to 6.00]

8. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) For Dextromethorphan and Dextrorphan on Cycle 2 Day 7
Description: Dextrorphan is an active metabolite of dextromethorphan.
Time Frame: Cycle 2 Day 7: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
hours
  Dextromethorphan | 3.00 [2.00 to 6.08]
  Dextrorphan | 4.00 [2.00 to 4.00]

9. Primary Outcome: Plasma Decay Half-Life (t1/2) For Dextrorphan 3 Days Prior to PF-00299804 Dosing
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Dextrorphan is an active metabolite of dextromethorphan.
Time Frame: Day -3: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
hours | 20.20 (28.645)

10. Primary Outcome: Plasma Decay Half-Life (t1/2) For Dextrorphan on Cycle 2 Day 7
Description: as for outcome 9
Time Frame: Cycle 2 Day 7: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
hours | 17.25 (15.935)

11. Primary Outcome: Oral Clearance For Dextromethorphan 3 Days Prior to PF-00299804 Dosing
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Day -3: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: Results not reported as data did not support calculation since levels of dextromethorphan were not tracked long enough for reliable estimation.
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 0

12. Primary Outcome: Oral Clearance For Dextromethorphan on Cycle 2 Day 7
Description: as for outcome 11
Time Frame: Cycle 2 Day 7: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 11
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 0

13. Primary Outcome: Urinary Metabolic Ratio (UMR) of Dextromethorphan to Dextrorphan 3 Days Prior to PF-00299804 Dosing
Description: The UMR was calculated as the ratio of the amount of dextrmotherphan excreted in urine from time zero to 8 hours post-dose on Day -3 to the amount of dextrorphan excreted in urine from time zero to 8 hours post-dose on Day -3.
Time Frame: 8 hours after dosing on Day -3
Population: PK parameter analysis population: all participants enrolled who were extensive metabolizers (EM), & treated who had at least 1 PK parameter of primary interest in at least 1 treatment period. EMs were defined as participants with a baseline UMR ≤0.3 & were either ultrarapid, extensive, or intermediate metabolizers as predicted by CYP2D6 genotyping.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 4
ratio | 0.008800 (0.017600)

14. Primary Outcome: Urinary Metabolic Ratio (UMR) of Dextromethorphan to Dextrorphan on Cycle 2 Day 7
Description: The UMR was calculated as the ratio of the amount of dextrmotherphan excreted in urine from time zero to 8 hours post-dose on Day 7 to the amount of dextrorphan excreted in urine from time zero to 8 hours post-dose on Day 7.
Time Frame: 8 hours after dosing on Day 7
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 5
ratio | 0.08040 (0.11042)

15. Secondary Outcome: Best Overall Response (BOR)
Description: BOR: investigator assessment by Response Evaluation Criteria in Solid Tumors (RECIST), recorded from treatment start until disease progression/recurrence. Complete Response: disappearance of all lesions. Partial Response (PR): >=30% decrease in sum of longest diameters (SLDs) of target lesions (TLs) taking as reference baseline SLD. Progressive disease (PD): >=20% increase in SLD of TLs taking as reference smallest SLD since treatment start, or appearance of >=1 new lesion. Stable disease: neither shrinkage for PR nor increase for PD taking as reference smallest SLD since treatment start.
Time Frame: Baseline, end of every even-numbered cycle until disease progression up to end of treatment (up to 18 months)
Population: Response anslysis set: all enrolled participants who received at least 1 dose of study medication and had an adequate baseline tumor assessment.
Measure: Number; unit: participants
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 7
participants
  Complete response | 0
  Partial response | 1
  Stable/No response | 1
  Objective progression | 5

16. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Baseline, end of every even-numbered cycle until disease progression up to end of treatment (up to 18 months)
Population: Participants with a response (CR or PR) in response analysis set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 1
weeks | NA [NA to NA] — One participant achieved partial response as best overall response on Day 42 and remained as partial response for the duration of the study. Therefore, data were not calculable.

17. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time in months from start of study treatment to first documentation of objective tumor progression or death due to cancer, whichever comes first. TTP was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.437. Tumor progression was determined from oncologic assessment data (where data meet the criteria for PD).
Time Frame: Baseline, end of every even-numbered cycle until disease progression up to end of treatment (up to 18 months)
Population: All enrolled participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 16
months | 1.4 [1.3 to NA] — Not calculable.

18. Other Pre Specified Outcome: Ratio of Dextromethorphan Area Under the Curve to Dextrorphan Area Under the Curve 3 Days Prior to PF-00299804 Dosing
Description: Dextrorphan is an active metabolite of dextromethorphan.
Time Frame: Day -3: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: Ratio of AUC was a derived parameter. As the primary endpoint for the study was not met, only the primary parameter AUC was analyzed and reported. Other parameters were not derived for this study based on investigator's decision.
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 0

19. Other Pre Specified Outcome: Ratio of Dextromethorphan Area Under the Curve to Dextrorphan Area Under the Curve on Cycle 2 Day 7
Description: Dextrorphan is an active metabolite of dextromethorphan.
Time Frame: Cycle 2 Day 7: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 18
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time that the participant provided informed consent through and including 28 calendar days after the last administration of the investigational product.
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-00299804 45 mg + Dextromethorphan 30 mg
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00299804 45 mg + Dextromethorphan 30 mg (N=15)
Colonic obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (General disorders) | 1
Chest pain (General disorders) | 1
Disease progression (General disorders) | 1
Pyelonephritis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00299804 45 mg + Dextromethorphan 30 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Deafness (Ear and labyrinth disorders) | 1
Ear disorder (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Oral pain (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Chest pain (General disorders) | 2
Early satiety (General disorders) | 1
Fatigue (General disorders) | 3
Mucosal inflammation (General disorders) | 5
Oedema (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Localised infection (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Seborroeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Dextromethorphan AUCinf and t1/2 results not reported as data did not support calculation since levels of dextromethorphan were not tracked long enough for reliable estimation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.